CLINICAL TRIAL: NCT03520673
Title: Primary Care Management of Lower Urinary Tract Symptoms in Men: Development and Validation of a Diagnostic and Clinical Decision Support Tool
Brief Title: Primary Care Management of Lower Urinary Tract Symptoms in Men
Acronym: PriMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPON 1553-16; 10327305 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2018-03-23; First posted 2018-05-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Primary Care; Urology
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Urodynamics

STUDY DESIGN:
Intervention Model Description: Diagnostic Accuracy Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Development of Clinical Decision Support Tool (Other): All men will receive the same series of simple index tests which will be compared with the results of the urodynamics reference test to identify which index tests give the best prediction of the urodynamic results. The data from the first cohort will develop the clinical decision support tool.
  Interventions: Diagnostic Test: Urodynamics

INTERVENTIONS:
Diagnostic Test: Urodynamics — All the men in the study will receive the urodynamics procedure as a reference test.

SUMMARY:
The PriMUS Study aims to develop a clinical decision support tool to help GPs more accurately diagnose and manage LUTS in men. The study will recruit 880 men across three research hubs in Bristol, Newcastle and Wales. Men will all receive a series of simple index tests in primary care (following NICE Clinical Guidelines) and a urodynamics reference test. The study will then compare which combination of the simple index tests give the best prediction of the urodynamics result, which can then be incorporated into the clinical decision support tool.

DETAILED DESCRIPTION:
Men are more likely to experience bothersome Lower Urinary Tract Symptoms (LUTS) as they get older. GPs follow standard processes to investigate signs of cancer, or more serious conditions but do not have access to tools to identify and manage more common symptoms of LUTS. This means men are likely to be referred to a urologist in secondary care, where they will receive advice or treatment that could have been given in primary care if GPs had more access to better diagnostic tools. The PriMUS Study will compare the results of the simple index tests, with the results of the urodynamic reference test, to identify which combination of simple index tests give the best prediction of the urodynamics diagnosis. The top performing simple index tests will be incorporated into the clinical decision support tool so that GPs can manage patients without needing invasive urodynamics. Follow up will be conducted 6 months post involvement; collating the treatment and management decisions made as a result of these procedures. The study will also consider and explore practicalities and acceptability of the urodynamic procedure and clinical decision support tool for both patients and clinical staff by conducting separate qualitative work.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 16 years and over.
* Men who present to their GP with a complaint of one or more bothersome lower urinary tract symptoms (LUTS)#
* Men able and willing to give informed consent for participation in study
* Men able and willing to undergo all index tests and reference test, and complete study documentation.

  * This would include men on current treatment, but who are still symptomatic

Exclusion criteria

* Men with neurological disease or injury affecting lower urinary tract function
* Men with LUTS considered secondary to current or past invasive treatment or radiotherapy for pelvic disease
* Men with other contraindications to urodynamics e.g. Heart valve or joint replacement surgery within the last 3 months, immunocompromised/immunosuppressed.
* Men with indwelling urinary catheters or who carry out intermittent self-catheterisation
* Men whose initial assessment suggests that clinical findings are suggestive of possible:

  * prostate or bladder cancer*
  * recurrent or persistent symptomatic UTI**
  * retention e.g. palpable bladder after voiding'
* Men unable to consent in English or Welsh where a suitable translator is not available. This is a multi-centre study based in primary care, and we cannot guarantee translation facilities at all sites

  * According to standard NHS cancer pathways. If later deemed unlikely, then eligible for study participation.

    * If UTI successfully treated but LUTS remain, then eligible for study

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 725 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Primary Outcome 1- Sensitivity and specificity of the PriMUS clinical decision aid in diagnosing detrusor underactivity, bladder outlet obstruction and detrusor over activity, in men with lower urinary tract symptoms presenting to primary care. | 36 months
  The accuracy of a clinical decision tool, which incorporates simple index tests, by reference and comparison to Urodynamic investigation as the gold standard at 36 months.

SECONDARY OUTCOMES:
Secondary Outcome 1 - Construction of a patient management algorithm to guide initial treatment for men with LUTS | 36 months
  Identify which combination of simple tests (including e.g. ethnicity, smoking status, height (cm) and weight (kg), medical history, medication, outcome of bladder diary, self-reported symptoms scores using IPSS and ICIQ questionnaires, Digital Rectal Examination Result, Prostate Specific Antigen (PSA) result, Abdominal Physical Examination Result) best predict the urodynamic diagnosis at 36 months.
Secondary Outcome 2 - Qualitative analysis of patients' and clinicians' views on the use of a LUTS decision aid in the primary care setting | 24 months
  Analyse the acceptability of a decision aid in primary care with patients and clinicians, to assess the decision tool's value and potential usability.
Secondary Outcome 3 - Estimate potential percentage change in referral rates to secondary care for men with LUTS | 36 months
  To calculate the potential change in referral rates of men with LUTs into secondary care to calculate the potential overall excess treatment cost savings.
Secondary Outcome 4 - Estimation of potential costs / savings of implementation of the primary care LUTS decision aid both from a population and individual patient perspective | 36 months
  Estimation of potential costs / savings of implementation of the primary care LUTS decision aid both from a population and individual patient perspective

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Edwards Profressor, Principal Investigator — Division of Population Medicine, Cardiff University; Chris Harding Mr, Principal Investigator — Newcastle Upon Tyne NHS Foundation Trust
Locations (1):
- Cardiff University, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No